CLINICAL TRIAL: NCT02841111
Title: Impact of Early Transfusions of Packed Red Cells on the Evolution of Renal Transplantation
Brief Title: Old Red Blood Cell In Renal Transplantation
Acronym: ORBIT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Agence de La Biomédecine (Other Government); Etablissement Français du Sang (Other); Amiens University Hospital (Other); University Hospital, Angers (Other Government); Bicetre Hospital (Other); University Hospital, Bordeaux (Other); University Hospital, Brest (Other); University Hospital, Caen (Other); University Hospital, Clermont-Ferrand (Other); CRC CHI Creteil France (Other Government); Centre Hospitalier Universitaire Dijon (Other); Hopital Foch (Other); University Hospital, Grenoble (Other); Groupe Hospitalier Pitie-Salpetriere (Other); University Hospital, Lille (Other); University Hospital, Limoges (Other); Hôpital Edouard Herriot (Other); Centre Hospitalier Lyon Sud (Other); University Hospital, Marseille (Other); University Hospital, Montpellier (Other); Central Hospital, Nancy, France (Other); Nantes University Hospital (Other); Hôpital Necker-Enfants Malades (Other); Centre Hospitalier Universitaire de Nice (Other); Poitiers University Hospital (Other); CHU de Reims (Other); Rennes University Hospital (Other); CHU de Rouen - Accueil (Other); Centre Hospitalier Universitaire de Saint Etienne (Other); Saint-Louis Hospital, Paris, France (Other); University Hospital, Strasbourg, France (Other); Tenon Hospital, Paris (Other); University Hospital, Toulouse (Other); University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: P/2013/166
Record Dates: First submitted 2016-07-19; First posted 2016-07-22 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Disorder Related to Renal Transplantation; Transfusion Reaction
MeSH Terms: conditions — Transfusion Reaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Kidney transplantation is the treatment of choice for ESRD. However, the life expectancy of kidney transplant patients is lower than that of the general population. Deaths recipients are due mainly to cardiovascular diseases related to a chronic inflammatory state. In addition, renal transplant patients frequently have anemia, identified as an independent cardiovascular risk factor that can be corrected by blood transfusion.

But the relationship between transfusion and inflammatory condition are bidirectional. The patient's inflammatory condition will sound on the effectiveness of transfusion and transfusion could trigger an inflammatory condition. This has been reported with the said blood components "aged", especially with packed red cells in patients hospitalized in intensive care after heavy heart surgery.The main objective of this study is to evaluate the impact of early transfusions on the evolution of renal transplantation (ie death, anti-HLA immunization, acute rejection, graft loss, delayed graft function, cardiovascular events ) taking into account in the analysis: patient age at the time of transplantation, the number of incompatibility (s) (HLA class I and / or II) between the graft and the patient and sex of the recipient.

This is a multicenter retrospective observational study (descriptive epidemiological study).The impact of early transfusions is determined retrospectively over a period of 6 years from 01 January 2002 to 31 December 2008, in renal transplant patients of all centers of France met the criteria for inclusion. This cohort represents about 12 000-14 000 patients

ELIGIBILITY:
Inclusion Criteria:

* male or female patients aged over 18 years
* patients who received a first kidney transplant

Exclusion Criteria:

* Patients who received multiple transplants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The impact of early transfusions is determined retrospectively over a period of 6 years from 01 January 2002 to 31 December 2008, in renal transplant patients of all centers of France met the criteria for inclusion. This cohort represents about 12 000-14 000 patients.
Sampling Method: Probability Sample
Enrollment: 12000 (Actual)
Dates: Start 2002-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
blood transfusion carried out within 14 days of transplantation (presence / absence) related to renal transplantation changes (i.e.: death, anti-HLA immunization, acute rejection, graft loss, delayed recovery of renal function, cardiovascular events) | 6 years

SECONDARY OUTCOMES:
blood transfusion carried out within 14 days of transplantation, taking into account the shelf life of CGR transfused, number of pockets transfused and the number of transfusion events related to renal transplantation changes. | 6 years

IPD SHARING:
Plan to Share IPD: No